CLINICAL TRIAL: NCT01318291
Title: An Assessment of the Effect of a Brief Psychological Intervention on Decreasing Drop-Out Rates in IVF Patients
Brief Title: Effect of Psychological Intervention on Drop-out Rates in IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston IVF (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alice D. Domar, PhD, Alice D. Domar, PhD, Boston IVF
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 38844
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Infertility
Keywords: IVF; Drop out
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Behavioral: Control
- CCRI Group (Experimental)
  Interventions: Behavioral: CCRI Group

INTERVENTIONS:
Behavioral: CCRI Group — Cognitive Coping and Relaxation Intervention (CCRI) Cognitive Coping and Relaxation Intervention (CCRI) group who will receive a packet of relaxation and stress management suggestions
  Arms: CCRI Group
Behavioral: Control — Medical treatment alone
  Arms: Control

SUMMARY:
The most common reason why insured In Vitro Fertilization (IVF) patients drop out of treatment is the distress caused by the treatment.

The objective of this study is to determine the efficacy of a combined Cognitive Coping and Relaxation Intervention (CCRI) in reducing drop out behavior in IVF patients.

DETAILED DESCRIPTION:
Intervention participants will be given a packet containing the CCRI, which consists of two intervention components tailored to the Stimulation Phase and Waiting Phases of IVF. The cognitive component of the CCRI is the PRCI intervention (Boivin & Lancastle, 2008) tailored to the stimulation/waiting phases of an IVF cycle. The PRCI intervention consists of a series of ten statements that facilitate the use of cognitive reappraisal coping, a form of coping that helps people think more about the positive aspects of a difficult situation and dwell less on problems or uncertainties of the future.

The relaxation components of the CCRI consists of techniques that have been used for two decades in the mind/body infertility program as well as in randomized controlled research trials. For the Stimulation phase, participants will receive instructions on how to do "mini relaxation" techniques which are specifically designed to reduce anxiety in the moment, for example feelings of tension, worry, and nervousness that might occur prior to and during Stimulation phase procedures (e.g. injections, blood tests, and ultrasounds). For the Waiting Phase the relaxation intervention will include a relaxation CD. The CD contains narrated instruction on how to elicit the relaxation response through several techniques

This is a randomized, controlled prospective study conducted at a private academically-affiliated infertility clinic and includes women ages 44 and below scheduled to undergo their first IVF cycle. Subjects are randomized to a CCRI or a control group. The primary outcome measure is dropout rates.

ELIGIBILITY:
Inclusion Criteria:

* First fresh IVF cycle
* Using own eggs
* Able to read, understand, and sign the informed consent in English
* Must have insurance coverage for IVF cycle

Exclusion Criteria:

* >1 previous IVF cycle
* Donor egg cycle

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Drop out rates | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alice D Domar, PhD, Principal Investigator — Boston IVF; Jacky Boivin, PhD, Study Director — School of Psychology, Cardiff University
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Domar AD, Gross J, Rooney K, Boivin J. Exploratory randomized trial on the effect of a brief psychological intervention on emotions, quality of life, discontinuation, and pregnancy rates in in vitro fertilization patients. Fertil Steril. 2015 Aug;104(2):440-51.e7. doi: 10.1016/j.fertnstert.2015.05.009. Epub 2015 Jun 13. PMID 26072382